CLINICAL TRIAL: NCT05886504
Title: DRIVE-Mind II (Drug Use & Infections in ViEtnam: Mental Health Intervention for INjecting Drug Users) Impact of Sustained Psychiatric Intervention for People Who Inject Drugs on Their Viral Exposure and Mental Health in Haiphong, Vietnam
Brief Title: Drug Use & Infections in ViEtnam: Mental Health Intervention for INjecting Drug Users
Acronym: DRIVEMINDII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Centre Pierre Nicole Croix-Rouge française (Unknown); Haiphong University of Medicine and Pharmacy (Other); Université Montpellier (Other); Center for supporting Community Developement Initiatives Hai Phong (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ANRS 0041s
Record Dates: First submitted 2023-05-10; First posted 2023-06-02 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Psychiatric Disorder; Drug Use
Keywords: psychosis; depression; suicidal risk; drug use; community-based psychiatric intervention
MeSH Terms: conditions — Mental Disorders; Psychotic Disorders; Depression

STUDY DESIGN:
Intervention Model Description: prospective cohort study comparing PWID diagnosed with a psychiatric disorder (depression, psychotic disorder, suicide risk) and getting benefit from a community-based psychiatric intervention to a control group of PWID free of psychiatric disorders. They will be mainly compared in terms of HIV/HCV exposure, severity of substance disorder, quality of life, sustainability of mental health improvement.
  Estimated enrolment: 600 participants (200 in the intervention group and 400 - 200 HIV-positive and 200 HIV-negative - in the control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychiatric intervention group (Active Comparator): 200 PWID diagnosed with either depression, psychosis or suicidal risk will be proposed to be included in the intervention arm Participants will receive free psychiatric consultation and medication on community-based organization (CBO) sites with full support from CBO members They will receive (together with the control group) linkage to care when needed (HIV, methadone treatment) and harm reduction services.
  Interventions: Other: Community-based psychiatric intervention
- control group free from psychiatric disorder (No Intervention): 200 PWID living with HIV and 200 PWID non-infected with HIV, both free of a diagnosis of depression, psychosis or suicidal risk, will be recruited and proposed a one year follow-up.
  They will receive (together with the intervention group) linkage to care when needed (HIV, methadone treatment) and harm reduction services.

INTERVENTIONS:
Other: Community-based psychiatric intervention — intervention will take place in CBO offices instead of mental health department, medication will be given freely and psychiatric consultations will be free. Trained CBO members will provide individual and collective support including recall of appointments and tracing of those lost to follow-up, information on mental health, main psychiatric disorders, psychiatric medication, their potential side effects and expected benefits, contact with families and continuous support
  Arms: Psychiatric intervention group

SUMMARY:
The main objective of this study is to show that People Who Inject Drugs (PWID) suffering initially from a major depressive disorder, a psychotic disorder and/or had a suicide risk and who received a community-based psychiatric intervention improve sustainably their mental health and are comparable after intervention to a population of PWID free of these disorders in terms of:

* HIV/HCV exposure
* Severity of substance use
* Quality of life This is prospective one-year cohort study comparing 200 PWID diagnosed with a psychiatric disorder with 400 controls (200 PWID living with HIV and 200 PWID non-infected with HIV, both free of a diagnosis of depression, psychosis, suicidal risk at cohort initiation).

Psychiatric intervention includes free psychiatric consultations and medications (issued on CBO sites), support from CBO members for appointments, information, treatment adherence, contact with families and tracing of those lost to follow-up. Target population and controls will also be proposed linkage to care (HIV, methadone) and harm reduction services.

ELIGIBILITY:
Inclusion Criteria:

Drive Mind II Psychiatric intervention group:

Participants of the ANRS 12353/National Institue of Drug Abuse (NIDA) Region of Interest (ROI) DA 041978 DRIVE study (age > 18 years; positive urine test for heroin and/or methamphetamine & skin marks of injection) who either:

* participated to the DRIVE Mind I cohort
* were candidate for the DM II control group but were diagnosed at inclusion with a major depressive disorder, psychotic disorder or suicide risk (MINI semi-structured interview) or any other significant psychiatric disorder requiring support and treatment (clinical diagnosis of a psychiatrist);
* participants recruited in the control group diagnosed at any step of the one-year follow-up with a major depressive disorder, a psychotic disorder or suicide risk (MINI semi-structured interview) or any other significant psychiatric disorder requiring support and treatment (clinical diagnosis of a psychiatrist) at M6 will be proposed to join the psychiatric cohort;
* Signed informed consent form. Participants eligible for the DM II cohort but refusing the principle of a treatment will nevertheless be included in the psychiatric cohort for follow-up, counselling and support except if the severity of the clinical situation requires immediate hospitalization in the mental health department.

Drive Mind II control group

Participants of the ANRS 12353/NIDA ROI DA 041978 DRIVE study (age > 18 years; positive urine test for heroin and/or methamphetamine & skin marks of injection):

* who participated to the DRIVE M30 survey and
* were screened negative for a potential psychiatric disorder at DRIVE M30 visit (Quick screening tool, QST) and
* are free of a major depressive disorder, a psychotic disorder or suicide risk (MINI semi-structured interview) or any other significant psychiatric disorder requiring support and treatment (clinical diagnosis of a psychiatrist) at DM II cohort initiation
* Signed informed consent form. Recruitment in the control group will take place until 200 HIV+ and 200 HIV- are enrolled

Exclusion Criteria:

* Severe psychiatric condition at cohort initiation requiring immediate hospitalization in the mental health department
* Severe associated diseases requiring specific treatment incompatible with a psychiatric ambulatory follow-up and treatment;
* Any condition which might, in the investigator's opinion, compromise the safety of the patient by participating in the study including very severe clinical condition;
* Contraindication for treatment with mirtazapine, sertraline, risperidone, olanzapine, sulpiride, quetiapine, melatonine;
* Person deprived of freedom by a judicial or administrative decision;
* Person who plan to move out from Hai Phong in the next 12 months;
* Person unable to understand the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Viral exposure score | Month 12
  Sum of the answers to several HIV/Hepatitis-C Virus (HCV)-related risk behaviors questions, weighed according to the significance of the risk (timeframe: last 6 months).
  Score range from 1 to 15. A higher score means a higher viral exposure
Severity of substance use score | Month 12
  Percentage of participants meeting at least one of the following criteria: persistent (last 6 months) injection practice (yes/no), daily heroin use (last 30 days), regular methamphetamine use (> 4 times/last 30 days), alcohol misuse (defined with audit-c questionnaire with score > 3 in men and > 2 in women during last 6 months).
  Score ranges from 1 to 4. Higher score means a higher severity of suubstance use.
  Each criteria will also be assessed individually.
Quality of life score | Month 12
  5 items and self-rated health evaluation of the EuroQol-5D Scale (Q5D-5L)

SECONDARY OUTCOMES:
Percentage of compliant participant :effectiveness of HIV treatment | Month 12
  HIV viral load among PWID living with HIV
Percentage of participant facing difficulty to access to care | Month 12
  Combination of quantitative and qualitative approaches will allow to quantify and describe structural or clinical factors conditioning access to care and which can explain the observed lack of therapeutics effectiveness in the population of the study.
Ppercentage of Psychiatric disorder associated with methamphetamine (meth) use | Month 12
  Incidence of methamphetamine-induced psychotic disorder, as measured by a clinical evaluation at each visit (using a MINI questionnaire plus clinical evaluation for confirmation)
HIV/HCV incidence | Month 12
  Comparaison of the incidence in the 2 arms
Incidence of psychiatric disorders in the control groups | Month 12
  Asessment for depression, psychosis and suicide risk at M0, M6 and M12 visits
Cost of a specialized community-based psychiatric intervention | Month 12
  Micro-costing analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Department, Haiphong, Hai Phong, Vietnam

IPD SHARING:
Plan to Share IPD: No